CLINICAL TRIAL: NCT03722082
Title: Study About the Effectiveness of Enhancing Cognitive Reserve in Children, Adolescents and Young Adults at Genetic Risk for Psychosis
Brief Title: Enhancing Cognitive Reserve of the Offsprings of Bipolar and Schizophrenic Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Clinic of Barcelona (Other)
Collaborators: Institut d'Investigacions Biomèdiques August Pi i Sunyer (Other); Consorcio Centro de Investigación Biomédica en Red (CIBER) (Other Government); Instituto de Salud Carlos III (Other Government)
Responsible Party: Principal Investigator, Carla Torrent, Principal Investigator, Hospital Clinic of Barcelona
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PI17/01066 and PI/1700741
Record Dates: First submitted 2018-10-11; First posted 2018-10-26 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-05

CONDITIONS: Bipolar and Related Disorders
Keywords: bipolar disorder; schizophrenia; offsprings
MeSH Terms: conditions — Bipolar and Related Disorders; Bipolar Disorder; Schizophrenia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Primary outcome
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhancing cognitive reserve intervention (Experimental): This intervention focuses in the improvement of academic skills, the increase of leisure activities and the improvement of neurocognitive functions with the ultimate goal of improving daily functioning. This intervention is based on ecological tasks that will be carried out in two areas, both in the hospital and at home. Most of the techniques are based on: pencil and paper tasks, with audiovisual and virtual reality support, telephone applications and group activities. The groups will be made with parents and children, adolescents and young adults separately being the content of the sessions the same but adapted to the age of the attendees.
  Interventions: Behavioral: Enhancing Cognitive Reserve
- Supportive Intervention (Placebo Comparator): The participants will not receive any structured intervention focused to enhance cognitive reserve. The therapists will adopt a client-centred focus, meaning that whatever problems the patient presents will be dealt with by providing emotional support and general advise.
  Interventions: Behavioral: Support intervention

INTERVENTIONS:
Behavioral: Enhancing Cognitive Reserve — The intervention is aimed at improving cognitive reserve in offsprings of patients diagnosed with schizophrenia or bipolar disorder. The program is composed of 12 sessions of 60 minutes and will be adapted according the three different age groups (6-12) (13-18) (18-25). Each group will include between 6-to-8 offsprings and conducted by 4 experienced neuropsychologists in both children and adults. The sessions are the following:
  Arms: Enhancing cognitive reserve intervention
Behavioral: Support intervention — The support group will schedule meetings with the participants in order to talk about their daily life with the possibility to talk about the difficulties they encounter.
  Arms: Supportive Intervention

SUMMARY:
The high hereditary component and the contribution of neurodevelopmental processes in bipolar disorder and schizophrenia means implies the children of these patients are considered a high risk population for both diseases and therefore a very adequate sample for the study of vulnerability markers to both disorders. To date there is no previous literature on the psychological approach of children and adolescents of bipolar or schizophrenic patients. The concept of cognitive reserve (CR) was initially developed in the field of dementia, it assumes that people with the same brain damage may have different clinical manifestations depending on their ability to compensate for this damage, so a greater cognitive reserve will entail a greater capacity to compensate the alterations and difficulties due to the pathology. Enhancing CR in high genetic risk population could help the acquisition of skills that help compensate the clinical, cognitive and neuroimaging alterations and ultimately help in the prevention of the development of pathologies for those with higher risk.This study aims to develop and apply a psychological program in order to enhance cognitive reserve (CR) in child, adolescent and young adults offspring of patients diagnosed with schizophrenia or bipolar disorder (SZBP-OFF).

DETAILED DESCRIPTION:
The project will have two main objectives: to test the effectiveness of the psychological program and to test if the observed improvements are stable over time (nine months of follow-up). A sample of 108 SZBP-OFF and 52 community controls will be included. Both groups will be assessed with clinical scales, neuropsychological, CR and neuroimaging assessments at baseline. Then, the SZBP-OFF group will be randomized to psychological program to enhance CR (N= 54) or to support treatment (N=54). SZBP-OFF subjects will be evaluated with clinical, CR, neuropsychological and neuroimaging tests after the psychological intervention and at nine months follow-up in order to assess if the obtained results are stable over time. The investigators hypothesize that SZBP-OFF will show lower CR scores and higher percentages of psychopathology, cognitive difficulties and brain abnormalities. The investigators also hypothesize that SZBP-OFF who received the psychological intervention will increase their CR and will decrease the severity of the observed difficulties (in clinical, neuropsychological, CR and neuroimaging areas). These results will be stable in the nine month follow-up assessment.

ELIGIBILITY:
Inclusion Criteria (Off-spring of patients) Inclusion criteria (Offsprings)

* Children, adolescents or young adults of both genders aged from 6 to 25, with the father and / or mother with schizophrenia, schizoaffective disorder or bipolar disorder according to DSM-IV criteria.
* Informed consent signed by their parents or legal guardians by adolescents if they are under 12 years old.

Inclusion criteria (Controls)

* Children, adolescents or young adults of both genders between the ages of 6 and 25 years.
* No history of psychotic disorder or bipolar disorder in first and second degree relatives.
* Consent signed by the parents or legal guardians if they are under 12 years old.

Exclusion Criteria:

• Mental retardation with impaired functioning and presence of neurological disorder or history of traumatic brain injury with loss of consciousness.

Ages: 6 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 173 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Cognitive reserve | 3 months afther the intervention and 12 months after baseline
  Changes in cognitive reserve assessed with a specific scale which assesses the most common proposed proxy indicators such as education-occupation' which is assessed taking into account the number of years of obligatory education that subjects completed and parent's educational level; and the lifetime school performance and lifetime participation in leisure, social and physical activities.

SECONDARY OUTCOMES:
Hamilton Depression Rating Scale (HDRS-21) | After the intervention (3 months) and 1 year after baseline
  Scale to assess depression symptoms. Score between 0 to 7 indicates absence of depressive symptoms, hihher scores indicate more severe depression.
Young Mania Rating Scale (YMRS) | After the intervention (3 months) and 1 year after baseline
  The YMRS is a rating scale used to evaluate manic symptoms at baseline and over time in individuals with mania. Scores superior to 12 indicate presence of manic episodes. Higher scores indicate more severe mania.
Bipolar Prodrome Symptom Interview and Scale_Prospective (BPSS_FP) | 12 months after baseline
  It is a specific interview for emerging bipolar disorder symptoms.
Continuous Performance Test | After the intervention (3 months) and 12 months after baseline
  Sustained attention test
Wisconsin Card Sorting Test | After the intervention (3 months) and 12 months after baseline
  Executive function test (set-shifting, flexibility)
Stroop Test | After the intervention (3 months) and 12 months after baseline
  Executive function test (inhibit interference)
Neuroimage variables | After the intervention (3 months)
  Changes in white and grey matter. Measure will be performed with a MRI

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clinic, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] de la Serna E, Montejo L, Sole B, Castro-Fornieles J, Camprodon-Boadas P, Sugranyes G, Rosa-Justicia M, Martinez-Aran A, Vieta E, Vicent-Gil M, Serra-Blasco M, Cardoner N, Torrent C. Effectiveness of enhancing cognitive reserve in children, adolescents and young adults at genetic risk for psychosis: Study protocol for a randomized controlled trial. Span J Psychiatry Ment Health. 2023 Jul-Sep;16(3):184-191. doi: 10.1016/j.rpsm.2021.02.003. Epub 2021 Feb 22. PMID 33631372